CLINICAL TRIAL: NCT06574581
Title: Allogenic Adipose Tissue Derived-MSCs Therapy in Patients With Connective Tissue Diseases-associated Interstitial Lung Disease(CTD-ILD): Phase I/IIa Clinical Trial
Brief Title: ADSCs Therapy in Patients With CTD-ILD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC1-042
Record Dates: First submitted 2024-08-01; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Connective Tissue Diseases; Interstitial Lung Disease
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADSC01 (Experimental): 1. Low-dose AD-MSC (1x10E6 cells/kg);
  2. Medium-dose AD-MSC (2x10E6 cells/kg)
  3. High-dose AD-MSC (3x10E6 cells/kg)
  Interventions: Biological: ADSC01

INTERVENTIONS:
Biological: ADSC01 — The initial 3 subjects will receive low-dose AD-MSC (1x10E6 cells/kg) infusion therapy only once; if no adverse events after 4 weeks, the next 4-7 subjects will receive medium-dose AD-MSC (1x10E6 cells/kg) infusion therapy twice; if no adverse events after 4 weeks of the last infusion, the next 8-10 subjects will receive high-dose AD-MSC (1x10E6 cells/kg) infusion therapy three times.

SUMMARY:
Connective tissue disease (CTD), an autoimmune and inflammatory disease, usually accompanied by lung interstitial/alveolar inflammation and fibrosis (so called interstitial lung disease, ILD). The prevalence and mortality rate of CTD-ILD increase in recent several years. Although the use of corticosteroids and strong immunosuppressants can improve ILD in some patients with CTD, progressive lung fibrosis which needs lung transplantation and results in respiratory failure, even with mortality is observed. Currently, stem cell therapy is a breakthrough in the treatment of CTD-ILD, and the effective therapy with stem cells for patients with ILD have been reported.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are adult multipotent cells with self-renewal capacity, and have immunomodulatory function. By virtue of these properties, they have an ability of tissues repairing as well as regeneration, and have immunomodulatory function through an interaction with immune cells. Compared with other MSCs, adipose tissue derived-MSC (AD-MSC) are attainable by a less invasive method, grow robustly, and have a high proliferation capacity and a low immunogenicity. Recently, AD-MSC is widely employed in the field of cardiovascular diseases and autoimmune diseases without the emergence of serious adverse events.

This is a Phase I/IIa, open-labelled (without placebo group) clinical trial to treat refractory or rapidly progressive ILD in 10 patients with CTD by intravenous transfusion with allogenic AD-MSC. After signing the informed consent, CTD-ILD patients will be enrolled in this trial, including pre-treatment evaluation, admission for intravenous transfusion with AD-MSC, and post-infusion follow-up. The initial 3 subjects will receive low-dose AD-MSC (1x10E6 cells/kg) infusion therapy only once; if no adverse events after 4 weeks, the next 4-7 subjects will receive AD-MSC (1x10E6 cells/kg) infusion therapy twice; if no adverse events after 4 weeks of the last infusion, the next 8-10 subjects will receive AD-MSC (1x10E6 cells/kg) infusion therapy three times. The major aims of this trial are to improve the outcome of CTD patients with refractory ILD or rapidly progressive ILD, and identify an optimal dose of the used AD-MSC

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged between 20 and 80 years who meet the diagnostic criteria for connective tissue diseases such as dermatomyositis, polymyositis, scleroderma, systemic lupus erythematosus, rheumatoid arthritis, or Sjogren's syndrome.
2. Subjects with refractory or progressive fibrotic interstitial lung disease: Subjects have been treated with steroids and potent immunosuppressants for more than 24 months with continued deterioration of lung function or lung lesions on CT scan (defined as a forced vital capacity (FVC) decline of more than 10% from baseline, an FVC decline of 5-10% with a diffusing capacity for carbon monoxide (DLCO) decline of more than 15% from baseline, or enlargement of lung lesions on CT scan) ; Or subjects with rapidly progressive interstitial lung disease: treated with high-dose steroids (above 0.8 mg/kg/day) and potent immunosuppressants for more than 3 months with continued deterioration of lung function or lung lesions on CT scan (defined as an FVC decline of more than 5% from baseline, a DLCO decline of more than 10% from baseline, or enlargement of lung lesions on CT scan); subjects with rapidly worsening condition: Onset of pulmonary symptoms within one month, gradual worsening of dyspnea and decreased blood oxygen levels, or enlargement of lung lesions.
3. Subjects must have a well-established family support system confirmed by interviews with the principal investigator and social worker.
4. Negative high-sensitivity urine pregnancy test before the trial.
5. Agree to use effective contraceptive measures during the trial (e.g., taking contraceptive pills or using intrauterine devices one month before the trial).

Exclusion Criteria:

1. Subjects who are unwilling to sign the informed consent form after detailed explanation by the physician.
2. Patients younger than 20 or older than 80 years who show improvement in lung function or lung lesions on CT scan after 6 months of treatment with steroids and immunosuppressants.
3. Women who are pregnant or breastfeeding, and women of childbearing age who do not use contraception.
4. Subjects with abnormal liver function (serum GOT and GPT levels more than twice the upper limit of 40 units, except those caused by inflammatory myopathy) or poor kidney function (serum creatinine levels exceeding 1.4 units).
5. Subjects with immune deficiencies such as HIV/AIDS or other specific conditions (e.g., those diagnosed with notifiable infectious diseases as per Ministry of Health announcements).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety profile (between the first infusion of AD-MSCs and 48 weeks after the last infusion of AD-MSCs) | 48 weeks
  1. Stable blood pressure: systolic pressure 90-120mmHg and diastolic pressure 60-80mmHg measured after resting for 10 minutes
  2. Stable pulse rate: ranges 60-100/minute after resting for 10 minutes
  3. Stable respiratory rate: ranges 12-20/minute after resting for 10 minutes
  4. Normal body temperature 35.7℃-37.9℃.
  5. Resting oxygen saturation≧90% without oxygen use.
  6. Absence of AD-MSCs infusion-related serious adverse event.

SECONDARY OUTCOMES:
Efficacy profile (between the first infusion of AD-MSCs and 48 weeks after the last infusion of AD-MSCs) | week 48.
  1. Change of six-minute walking distance(6MWD): Increase of 6MWD≧5% from baseline at week 12, 8% at week 24, 10% at week 48.
  2. St. George's Respiratory Questionnaire: Change of score≧5% from baseline at week 12, 10% at week 24, 15% at week 48.
  3. Quality of life (SF-36): Increase of score≧5% from baseline at week 12, 8% at week 24, 10% at week 48.
  4. Forced vital capacity (FVC): Decrement of FVC<5% at week 12, increment ≧5% at week 24, increment ≧10% at week 48.
  5. Diffusing capacity for carbon monoxide (DLco): Decrement of DLco <5% at week 12, increment≧5% at week 24, increment≧10% at week 48
  6. The extent of ILD (interstitial lung disease) lesion in HRCT: Decrement of ILD extent≧5% at week 24, and decrement of ILD extent≧10% at week 48.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan